CLINICAL TRIAL: NCT06720857
Title: Predictive Value of SFlt-1/PlGF Ratio for the Diagnosis of Cardiovascular Disorders in the Puerperium: Pilot Study
Acronym: SOMP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOMP
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Disorder; Puerperium; Disease
Keywords: SFlt-1/PlGF ratio
MeSH Terms: conditions — Cardiovascular Diseases; Puerperal Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypertensive disorders in the puerperium (Experimental): Identification of a risk stratification model and its predictive value for cardiovascular disorders in the puerperium
  Interventions: Diagnostic Test: Identification of a risk stratification model and its predictive value for cardiovascular disorders in the puerperium

INTERVENTIONS:
Diagnostic Test: Identification of a risk stratification model and its predictive value for cardiovascular disorders in the puerperium — Identification of a risk stratification model for cardiovascular/hypertensive disorders in the puerperium using a panel of placental biochemical markers (sFlt-1 and PlGF: already used in pregnancy for prediction of preeclampsia), demographic, clinical and laboratory data.

SUMMARY:
The goal of this clinical trial is to identify a risk stratification model and its predictive value for cardiovascular/hypertensive disorders in the puerperium (6 weeks postpartum) by making use of a panel of placental biochemical markers (sFlt-1 and PlGF: already used in pregnancy for prediction of preeclampsia), demographic, clinical and laboratory data. The goal is to create a score that allows the clinician to identify those expectant mothers who at discharge are at increased risk of developing cardiovascular/hypertensive disorders.

DETAILED DESCRIPTION:
At the time of recruitment, patients will be adequately informed about the purpose and modality of the study and will sign an informed consent form for participation in the study. On the first postpartum day, on the occasion of the blood tests included in the normal care routine, the patients will undergo measurement of circulating levels of angiogenic factors (soluble fms-like tyrosine kinase, sFlt-1; placental growth factor, PlGF), already used in pregnancy for predicting the risk of early and late preeclampsia. Marker assay kits will be provided free of charge by the company DASIT. Prior to collection, systolic and diastolic blood pressure will be measured by manual sphygmomanometer in supine position after at least 15 minutes of rest.

Anamnestic, clinical and laboratory data regarding pregnancy, childbirth and puerperium will be collected.

A diary for recording blood pressure values in the puerperium will be provided on the same occasion. The patient will be instructed in home blood pressure monitoring which should take place twice a week for the next 6 weeks after delivery. Return of the diary containing the pressure data will be done by e-mail. Postpartum hypertension is defined according to ACOG criteria as a systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg. If altered blood pressure values are found, the patient will be invited to go to the emergency department or to her primary care physician and treated according the usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 44 years
* Single pregnancy
* Understanding and obtaining informed consent

Exclusion Criteria:

* Language misunderstanding
* Twin pregnancies
* Inability to comply with study arrangements (e.g., inability to home recording of blood pressure values)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of a risk stratification model and its predictive value for cardiovascular/hypertensive disorders in the puerperium (6 weeks after delivery) | "From enrollment to the end of treatment (6 weeks after delivery)
  Through a panel of placental biochemical markers (sFlt-1 and PlGF: already used in pregnancy to predict preeclampsia), demographic, clinical and laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Farina, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy